CLINICAL TRIAL: NCT00222547
Title: Deworming and Enhanced Vitamin A Supplementation DEVTA Project
Brief Title: Deworming and Enhanced Vitamin A Every 6 Month in Rural Indian Children Aged 1-6
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: DEVTA
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2005-10-28 (Estimated); Status verified 2005-02

CONDITIONS: Village Children
MeSH Terms: interventions — Vitamin A; Albendazole

INTERVENTIONS:
Drug: Vitamin A
Drug: Albendazole

SUMMARY:
Randomisation of 72 large rural areas ("blocks") into a 2 x 2 trial of six- monthly treatment of all village children aged 1-5 with albendazole(400mg), vitamin A (200000 iu), both or neither. The placebo group get no trial treatment at all and do not receive physical placebos.

ELIGIBILITY:
InclusionCriteria:

* Area of residence

Exclusion Criteria:

* NONE

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 720000
Dates: Start 1999-01; Study Completion 2005-02

PRIMARY OUTCOMES:
childhood mortality rate at age 1-6

SECONDARY OUTCOMES:
fecal egg counts, plasma retinal, growth, sign of Vitamin A deficiency

CONTACTS AND LOCATIONS:
Overall Officials: Shally Awasthi, MD, Study Chair — King George Medical University, Lucknow
Locations (1):
- Shally Awasthi, Lucknow, Uttar Pradesh, India

REFERENCES:
- [Derived] Awasthi S, Peto R, Read S, Richards SM, Pande V, Bundy D; DEVTA (Deworming and Enhanced Vitamin A) team. Population deworming every 6 months with albendazole in 1 million pre-school children in North India: DEVTA, a cluster-randomised trial. Lancet. 2013 Apr 27;381(9876):1478-86. doi: 10.1016/S0140-6736(12)62126-6. Epub 2013 Mar 14. PMID 23498850
- [Derived] Awasthi S, Peto R, Read S, Clark S, Pande V, Bundy D; DEVTA (Deworming and Enhanced Vitamin A) team. Vitamin A supplementation every 6 months with retinol in 1 million pre-school children in north India: DEVTA, a cluster-randomised trial. Lancet. 2013 Apr 27;381(9876):1469-77. doi: 10.1016/S0140-6736(12)62125-4. Epub 2013 Mar 14. PMID 23498849